CLINICAL TRIAL: NCT02323477
Title: The Efficacy and Safety Assessment of Human Umbilical Cord Stroma-derived Multipotent Stromal Cells in Myocardial Infarction; a Phase 1/2 Clinical Trial (HUC-HEART Study)
Brief Title: Human Umbilical Cord Stroma MSC in Myocardial Infarction
Acronym: HUC-HEART
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to budget limitations as allocated for a given period.
Sponsor: Ankara University (Other)
Collaborators: Hacettepe University (Other); Turkiye Yuksek Ihtisas Education and Research Hospital (Other Government); Atigen-Cell and Tissue Center (Industry); Dr. Sami Ulus Children's Hospital (Other); Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Alp Can, Prof. Dr., Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 741.STZ.2014
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Chronic Ischemic Cardiomyopathy; Coronary Artery Bypass Surgery
Keywords: cellular therapy; chronic ischemic heart disease; phase 1/2 clinical study; human umbilical cord multipotent stem cell; human umbilical cord mesenchymal stem cell; ischemic heart disease; bone marrow mononuclear cell; allogeneic stem cell transplantation
MeSH Terms: conditions — Myocardial Ischemia | interventions — Stem Cell Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Allogeneic umbilical cord MSC group (Experimental): Allogeneic human umbilical cord MSCs will be transplanted to 39 male patients (age 30-80) intramyocardially during CABG in chronic ischemic cardiomyopathy (EF<%45)
  Interventions: Biological: stem cell transplantation
- Autologous bone marrow-derived MNC group (Active Comparator): Autologous bone marrow-derived MNCs will be transplanted to 20 male patients (age 30-80) intramyocardially during CABG in chronic ischemic cardiomyopathy (EF<%45)
  Interventions: Biological: stem cell transplantation
- Control group (No Intervention): 20 male patients (age 30-80) undergoing CABG in chronic ischemic cardiomyopathy (EF<%45) whom will not received any further transplantation

INTERVENTIONS:
Biological: stem cell transplantation — Human allogeneic umbilical cord MSC or autologous BM-MNC transplantation
  Arms: Allogeneic umbilical cord MSC group; Autologous bone marrow-derived MNC group

SUMMARY:
The purpose of this phase 1/2 clinical trial is to evaluate the efficacy and safety of allogeneic human umbilical cordstroma derived multipotent stem cells (hUCS-MSCs) in myocardial infarction (MI). All subjects will be taken into the bypass coronary surgery prior to the cell administration. This 2-year study comprise three independent groups, where the first group (n=20) will take no cells, second group will take autologous BM-MNCs (n=20), and third group (n=39) will be receiving allogeneic hUCS-MSCs. In all transplantations cells will be administered to the approximately 10 peri-infarct areas at one time. The infarct zone will be determined by the MR, SPECT and PET imaging. Only male subjects between 30-80 years of age. The efficiency of the therapy will be evaluated according to the parameters measured by MR, SPECT, and Echocardiography. All subject were taken into those measurements prior and 6, 12, 18 and 24 months after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic hearth disease who will experience CABG
* %25<EF<%45
* NYHA class II-IV patients
* hemodynamically stable

Exclusion Criteria:

* Patient's in approval
* Acute cardiac decompensation
* Acute myocardial infarction
* Congenital heart disease
* Additional surgical heart disease other than coronary artery disease
* Malign arrhythmia
* All malignancies
* HbA1c level >%10 (86 mmol/mol) type II diabetes mellitus
* Severe liver dysfunction
* Severe COPD
* Coagulopathy
* Immunosuppressive treatment
* Acute hepatitis, hepatitis B, C and HIV infection
* Chronic liver and renal failure
* Collagen tissue disease
* Stroke
* TB
* Hematological diseases
* Socially and mentally disabilities

Ages: 30 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
ventricular remodeling | within one year after cell transplantation
  Outcome measures will be determined by cardiac MR, SPECT and PET monitoring to assess the left ventricular ejection fraction (%), left ventricle end-diastolic and end-systolic volumes (mL/m2), left ventricle mass (g/m2), infarct size (%), and the thickness of the dysfunctional wall (mm).

CONTACTS AND LOCATIONS:
Locations (1):
- Alp Can, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Ulus AT, Mungan C, Kurtoglu M, Celikkan FT, Akyol M, Sucu M, Toru M, Gul SS, Cinar O, Can A. Intramyocardial Transplantation of Umbilical Cord Mesenchymal Stromal Cells in Chronic Ischemic Cardiomyopathy: A Controlled, Randomized Clinical Trial (HUC-HEART Trial). Int J Stem Cells. 2020 Nov 30;13(3):364-376. doi: 10.15283/ijsc20075. PMID 32840230
- [Derived] Can A, Ulus AT, Cinar O, Topal Celikkan F, Simsek E, Akyol M, Canpolat U, Erturk M, Kara F, Ilhan O. Human Umbilical Cord Mesenchymal Stromal Cell Transplantation in Myocardial Ischemia (HUC-HEART Trial). A Study Protocol of a Phase 1/2, Controlled and Randomized Trial in Combination with Coronary Artery Bypass Grafting. Stem Cell Rev Rep. 2015 Oct;11(5):752-60. doi: 10.1007/s12015-015-9601-0. PMID 26123356